CLINICAL TRIAL: NCT05863000
Title: Patient Behavior in Region H: How Does Illness Affect How You Act and Master Your Life?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anette Lykke Hindhede, Senior researcher, Associate professor, Rigshospitalet, Denmark
Other Study IDs: P-2022-764
Record Dates: First submitted 2023-05-04; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Comparison, Social
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in Region H: The health care system in Region H consists of 10 hospitals, including Region H's Psychiatry which consists of 11 centers. The hospitals annually have around 3 million visits from outpatients
  Interventions: Other: Online questionnaire/survey

INTERVENTIONS:
Other: Online questionnaire/survey — Participants are expected to answer a short survey based on their overall experiences with their own health. No participants will therefore be followed for more than the duration of time it takes a subject to answer the questionnaire (approx 15 minutes). Randomly selected volunteers of around 30 respondents will afterwards be invited to participate in a qualitative interview with the intend to elaborate their questionnaire responds.

SUMMARY:
This study investigates how the behavior within different patient groups are affected differently by illness and disease. The investigators ask how participants experience and approach their own health in order to gain insight on the implications of illness and disease on the individual's everyday life and how participants act and think regarding their own health and wellbeing across different patient groups. The investigators' hypothesis is that illness and disease is experienced as a great disturbance and an actor of change in a person's everyday life. Each person has their own individual experience and reaction to this disturbance. Still, there is less evidence for how disparate resources and socioeconomic statuses shape how patients react to this great change in their lives. Here the investigators expect to find demographic patterns across patient groups. The study carries a quantitative and qualitative approach with a broad target population which includes both patients with acute or chronic, serious, or less serious, somatic as well as psychiatric illnesses. The study is placed within the academic traditions of sociological health and disease mapping.

ELIGIBILITY:
Inclusion Criteria:

* The patient is assigned to Region H
* The patient is over the age of 18
* The patient is able to answer the questions

Exclusion Criteria:

* - The patient refuses to give informed consent
* The patient doesn't speak danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population consists of patients connected to a hospital clinic in Region H. We aim for a representative sample of patients in general and specific patient groups connected to a hospital within Region Hovedstaden
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Online questionnaire/survey | six months
  Investigators have developed a medical education survey in Danish for the participants to answer individually or with investigators' help. Participants are expected to give their informed consent before beginning the survey. In order to verify the quality of the survey investigators conducted preliminary cognitive interviewing on 10 participants broadly represented by gender, age, diagnosis' etc. Cognitive interviewing is an evidence based qualitative research method designed to investigate if a questionnaire fulfills its intended purpose and thereby ensures to improve education surveys . With help from an investigator respondents are expected to "think out loud" while answering the questionnaire. In the questionnaire, investigators ask participants about their socioeconomic background as well as questions about exercise, diets, alcohol, mental well being often in the context of their actions before and after receiving a diagnosis or becoming ill.

SECONDARY OUTCOMES:
Multiple correspondence analysis | through study completion, an average of 6 months
  Investigators plan to interpret investigators' data through a Multiple Correspondence Analysis (MCA) . MCA is a statistical approach utilized among others by sociologist Pierre Bourdieu in order to construct social fields and spaces with his empirical data . Through MCA investigators can analyze the pattern of relationships of several categorical dependent variables such as diagnosis, income, age, diet, geography etc.
  As such, it can also be seen as a generalization of principal component analysis when the variables to be analyzed are categorical instead of quantitative

CONTACTS AND LOCATIONS:
Locations (1):
- Anette Lykke Hindhede, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No